CLINICAL TRIAL: NCT04704648
Title: Feasibility Study of Ocular Surface Squamous Neoplasia (OSSN) Surgical Excision in People Living With HIV in Sub-Saharan Africa (SSA)
Brief Title: Feasibility Study of Ocular Surface Squamous Neoplasia Surgical Excision in People Living With HIV in Sub-Saharan Africa
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Retraining on study procedures required
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-104; UM1CA121947 (NIH)
Record Dates: First submitted 2020-11-30; First posted 2021-01-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Ocular Surface Squamous Neoplasia; HPV
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Using an exact binomial one-sample test for proportions, 90% power and one-sided 0.0167 significance level (0.05/3 = 0.0167), the number of study participants required to test the hypotheses shown above, respectively, are 28, 28 and 68. Thus, this study will require 68 evaluable participants using a one-sample test of proportions. We define evaluable as participants with suspected OSSN lesions who are shown to have OSSN on biopsy. We estimate that 20% of participants will be found to have lesions that are histopathologically not OSSN and will therefore, not be evaluable. As a result, we are recruiting 84 individuals (21 per clinical site) to get 68 evaluable participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Excision (Other): Treatment involves EXCISION ONLY (surgery) for the conjunctival lesion with 3 mm margins. Surgeons (registered as investigators at each site) will perform the operation in accordance with the procedures outlined in the AMC-104 manual of procedures (MOP). Standard of care topical antibiotics are given for infection prevention following surgery. No drugs or device treatments are administered for treatment of OSSN in this protocol.
  Interventions: Procedure: Surgical

INTERVENTIONS:
Procedure: Surgical — The treatment involves excision only of the conjunctival lesion with 3 mm margins. Surgeons (registered as investigators at each site) will perform the operation in accordance with the procedures outlined in the AMC-104 manual of procedures (MOP).
  As part of the study patients will be asked to return for follow-up evaluation 1 week, 6 weeks, 6 months, and 12 months after surgery. At each of these follow-up visits, the AMC-certified ophthalmologist will obtain a thorough ocular history as well as a history of AIDS-defining illnesses and perform a slit-lamp examination of both eyes, complete with templated drawings of the conjunctiva, and careful examination of the cornea for limbal stem cell deficiency.

SUMMARY:
Participants will undergo surgical excision of OSSN at baseline and will be followed at 1 week, 6 weeks, 6 months, and 12 months for post-surgical follow up. This study is being conduced to assess the feasibility of conducting multi-center prospective studies on surgical excision of suspected OSSN lesions in SSA in people living with HIV/AIDS (PLWHA). Participants include those with HIV infection and with suspected non-invasive OSSN lesions that the AMC-certified ophthalmologist determines can be resected with 3 mm clinical margins, sparing involvement of the superior and inferior fornices and 6 clock hours of the corneal scleral limbus.

DETAILED DESCRIPTION:
The AMC-certified ophthalmologist will obtain a thorough eye history and conduct a slit-lamp examination of both eyes. The AMC-certified ophthalmologist will draw the size and shape of the suspected lesion on a well-accepted template designed for documentation of ocular surface malignancies. Using this template, the AMC-certified ophthalmologist will document the number of clock hours of corneal-scleral limbus involved (6 clock hours maximum) as well as the maximum vertical and horizontal dimensions of the lesion in mm as determined through the use of the adjustable slit beam, whose length can be adjusted and determined using the slit length display window, a standard feature of slit lamp biomicroscopes.

Eighty-four participants undergoing surgical excision of tumors suspicious for OSSN will be enrolled in this study. Participants who do not complete the study follow-up visits will not be replaced. The lesions will be swabbed prior to surgical excision and the swabs will be placed in PrimeStore MTM solution, for HPV DNA testing. The suspected OSSN lesion will be excised with 3 mm margins as determined by clinical exam. The PrimeStore MTM solution will be sent to Stellenbosch University in Cape Town, South Africa for HPV testing. The surgically excised lesions will be fixed, aligned, embedded in paraffin, sectioned and evaluated by pathologists at each of the 4 study sites. Tissue will then be sent to Stellenbosch University in Cape Town, South Africa for confirmatory histopathologic analysis and HPV testing.

To ensure reliable follow-up, we will collect detailed contact and alternate contact information from study participants. Participants will be asked to return for follow-up one week after surgery, 6 weeks after surgery, 6 months after surgery, and 12 months after surgery. At each of these follow-up visits, the AMC-certified ophthalmologist will obtain a thorough medical history and perform a slit-lamp examination of the eyes. At week 2, sites will contact participants via phone to review AEs. Participants will undergo a structured review of post-surgical signs and symptoms at each follow-up visit. Participants presenting with a suspected recurrent OSSN lesion at follow-up will undergo re-excision per routine clinical care, including any follow-up per the local standard of care. After local diagnostic review, excised specimens will be sent for central histopathology evaluation and confirmation of recurrent OSSN or not recurrent OSSN. All other ocular lesions and conditions will be referred for routine medical care, outside of the study.

ELIGIBILITY:
Inclusion Criteria:

3.2.1 Participants with suspected unilateral, non-invasive OSSN lesions that the AMC-certified ophthalmologist determines can be resected with 3 mm clinical margins, sparing involvement of the superior and inferior fornices as well as 6 clock hours of the corneal scleral limbus. This assessment must be carried out within 4 weeks before surgery.

3.2.2 HIV positive. Documentation of HIV-1 infection by means of any one of the following:

* Documentation of receipt of ART by a licensed health care provider (Documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name. Antiretroviral drug regimens used for pre-exposure prophylaxis (PrEP) may not satisfy this requirement.;
* HIV-1 RNA detection by a licensed HIV-1 RNA assay demonstrating >1000 RNA copies/mL confirmed by a licensed screening antibody and/or HIV antibody/antigen combination assay;
* Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay.

Note: The term "licensed" refers to a kit that has been certified or licensed by an oversight body within the participating country and validated internally (e.g., U.S. FDA).

WHO and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an enzyme or chemiluminescence assay (E/CIA) that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

3.2.3 Performance status ≤ 2 on the WHO Scale (see Appendix III).

Exclusion Criteria:

3.3.1 Participants who are receiving any other investigational agents within 30 days before enrollment for surgery, except for investigational ART regimens, which will be permitted.

3.3.2 Participants with known history of ocular surface lesions including OSSN, other ocular neoplasm, pterygia, or limbal vernal keratoconjunctivitis.

3.3.3 Uncontrolled intercurrent illness within 4 weeks before enrollment, including but not limited to ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of 3 feasibility criteria across all participants and satisfaction of the feasibility criteria by at least 3 of 4 of the participating centers | 12 months
  * Slides from excised suspected OSSN lesions are successfully reviewed by central pathology and results of histopathology are communicated with the original site (i.e., meet all four criteria noted above) (Null hypothesis: p=0.5 vs. Alternative hypothesis: p≥0.8).
  * Participants undergoing suspected OSSN excision will not develop serious complications as defined in Section 4.4 (Observed complication rate of less than 20%).
  * Participants with biopsy-proven OSSN return for follow-up at 12 months (Null hypothesis: p=0.5 vs. Alternative hypothesis: p≥0.7).

SECONDARY OUTCOMES:
Proportion of participants with suspected OSSN lesions who are found to have biopsy-proven OSSN. | 12 months
  Participants presenting with a suspected recurrent OSSN lesion at follow-up will undergo re-excision per routine clinical care, including any follow-up per the local standard of care. After local diagnostic review, excised specimens will be sent for central histopathology evaluation and confirmation of recurrent OSSN or not recurrent OSSN.
To estimate the proportion of biopsy-proven OSSN lesions excised with clear margins on histopathologic analysis. | 12 months
  Participants presenting with a suspected recurrent OSSN lesion at follow-up will undergo re-excision per routine clinical care, including any follow-up per the local standard of care. After local diagnostic review, excised specimens will be sent for central histopathology evaluation and confirmation of recurrent OSSN or not recurrent OSSN.
To characterize the nature and frequency of surgical complications in participants undergoing excision of suspected OSSN. | 12 months
  The chi-square test without continuity correction will be used to compare the sites. If a significant difference between sites is detected with respect to any of the feasibility endpoints.
  • Do not develop surgical complications.
To estimate 1-year recurrence rates of biopsy-proven OSSN following surgical excision. | 12 months
  We will use the HybriSpot HPV Direct Flow Chip kit (Master Diagnóstica) to detect HPV DNA in formalin-fixed paraffin-embedded (FFPE) tissue samples.
To determine whether HPV is present in biopsy-proven OSSN pathology specimens. | 12 months
  We will use the HybriSpot HPV Direct Flow Chip kit (Master Diagnóstica) to detect HPV DNA in formalin-fixed paraffin-embedded (FFPE) tissue samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Uganda Cancer Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No